CLINICAL TRIAL: NCT02080143
Title: A Randomized, Open-Label, Comparative Study To Evaluate the Adhesion and Temperature Properties of Two Air-Activated, Adhesive Backed Heat Patches in Healthy Volunteers
Brief Title: A Comparative Study to Evaluate Two Air-Activated Adhesive Backed Heat Patches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Chattem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014003
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Skin temperature measurements; Heat patch adhesion; Dermal irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air Activated Heat Patch (Experimental): The experimental air activated heat patch will be worn by the subjects for 8 hours.
  Interventions: Device: Thermal Adhesion Patch
- Marketed ThermaCare Air Activated Heat Patch (Active Comparator): The marketed air activated heat patch will be worn by the subjects for 8 hours.
  Interventions: Device: Thermal Adhesion Patch

INTERVENTIONS:
Device: Thermal Adhesion Patch
  Other Names: Experimental Adhesion Patch
  Arms: Air Activated Heat Patch
Device: Thermal Adhesion Patch
  Other Names: Marketed ThermaCare Thermal Adhesion Patch
  Arms: Marketed ThermaCare Air Activated Heat Patch

SUMMARY:
A disposable, air-activated, adhesive backed heat patch is being evaluated.

Study terminated -O subjects.

DETAILED DESCRIPTION:
Study Protocol Terminated--0 subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects who complete an appropriately administered informed consent process that includes signing the IRB-approved consent form;
* subjects 18-75 years old of each sex;
* are of any skin type or race, providing the skin pigmentation will allow discernment of erythema;
* subjects who are in good general health and free of any disease state or physical condition;
* subjects who are willing and able to have the study products applied as directed, and comply with study instructions;
* subjects must be willing to restrict their activity for the 8 hour patch wear time so that patches and thermocouples do not come loose;
* subjects must be willing to wear a pouch containing the thermologger and thermocouple wiring for the entire 8 hours;
* subjects who are 55 years or older agree to wear a t-shirt provided by the site for the entire 8 hour patch wear time.

Exclusion Criteria:

* Subjects who are pregnant or nursing;
* subjects with excessive hair at the application site, scar tissue, tattoo or coloration that would interfere with the placement of the study product or the skin assessment;
* subjects with diabetes or poor circulation or have any clinically significant chronic illness which could place the subject at increased risk during participation or result in inappropriate dermal response during the study;
* subjects unable to feel pain or heat (e.g., subjects with neuropathy);
* subjects with active dermatitis (including sunburn) in the treatment area or other visible dermatological disease which, in the investigator's opinion, might interfere with the response to the study products or interfere with the skin assessments associated with the study products;
* have history of significant dermatologic cancers or neoplasms in the treatment area;
* subjects who have used topical dermatological products in the application area within 24 hours prior to anticipated study product application;
* subjects using a concomitant medication that, in the investigator's opinion, could interfere with the interpretation of the study results. Examples of such drugs include vasoactive (constrictor or dilator) medications, prescription or OTC, that could modulate blood flow, within 24 hours prior to or during the application of study products, including nitroglycerin, non-steroidal anti-inflammatory products (NSAIDs, e.g., ibuprofen, aspirin (<=81 mg/day is acceptable)), topical corticosteroids and OTC cough/cold products including antihistamines and/or either phenylpropanolamine or phentolamine;
* subjects who have used systemic steroids (i.e., oral, IV, IM or intra-articular) 30 days prior to the application of test articles (intranasal/inhaled steroids are acceptable);
* subjects who have received an investigational medication or device within 30 days prior to enrollment into this study;
* subjects who have a history of sensitivity to any of the study products or adhesion materials;
* subjects who are currently participating in an investigational study;
* subjects who are known to be noncompliant or are unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, product dependency, mental incapacity) in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Heat Intensity | 8 hours
  Assessed using sensors.

SECONDARY OUTCOMES:
Adhesion Evaluation | 8 hours
  Adhesion will be evaluated by visual assessment.
Irritation Evaluation | 8 hours
  At the conclusion of the study and upon removal of the heat patch the application area will be observed by a trained skin grader for visual signs of irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Q. Tejada, MD, Principal Investigator — Radiant Research, Inc.
Locations (1):
- Radiant Research, Inc., Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: No